CLINICAL TRIAL: NCT00329849
Title: A Phase 3, Randomized, Observer-blind, Controlled, Multi-Center Study to Compare the Safety of One Dose of Novartis Meningococcal ACWY Conjugate Vaccine With That of a Licensed Meningococcal ACWY Polysaccharide Vaccine (Menomune®) Administered to Healthy Children 2 to 10 Years of Age
Brief Title: Safety and Immunogenicity of Meningococcal ACWY Conjugate Versus Polysaccharide Vaccine in Children 2 to 10 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V59P10
Record Dates: First submitted 2006-05-23; First posted 2006-05-25 (Estimated); Results first posted 2013-11-05 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Meningococcal Disease
Keywords: Meningitis; children; vaccine; safety; efficacy
MeSH Terms: conditions — Meningococcal Infections; Meningitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- MenACWY-CRM (Experimental): Subjects ≥2 to ≤10 years of age received one dose of a quadrivalent meningococcal conjugate vaccine (MenACWY-CRM)
  Interventions: Biological: Meningococcal ACWY-CRM conjugate vaccine
- MenACWY-PS (Active Comparator): Subjects ≥2 to ≤10 years of age received one dose of a quadrivalent meningococcal polysaccharide (PS) vaccine (MenACWY-PS)
  Interventions: Biological: Meningococcal ACWY-PS polysaccharide vaccine

INTERVENTIONS:
Biological: Meningococcal ACWY-CRM conjugate vaccine — MenACWY-CRM vaccine was obtained by extemporaneous mixing of the lyophilized MenA component to be resuspended with the liquid MenCWY component. One dose (0.5 mL) was administered by IM injection in the deltoid area of the arm without a BCG scar.
  Arms: MenACWY-CRM
Biological: Meningococcal ACWY-PS polysaccharide vaccine — MenACWY-PS vaccine was supplied as a single dose (one vial of vaccine and one vial of diluent). One dose (0.5 mL) of MenACWY-PS vaccine was administered by SC injection in the deltoid area of the arm without a BCG scar.
  Arms: MenACWY-PS

SUMMARY:
Safety and immunogenicity of meningococcal ACWY conjugate versus polysaccharide vaccine in children 2 to 10 years of age

ELIGIBILITY:
Inclusion Criteria:

* Healthy children 2 to 10 years of age inclusive whose parents or legal guardians gave written informed consent at the time of enrollment;
* Available for all visits and telephone calls (parents or legal guardians) scheduled for the study;
* Good health as determined by the clinical judgment of the investigator.

Exclusion Criteria:

Individuals not eligible to be enrolled into the study were those:

* whose parent or legal guardian was unwilling or unable to give written informed consent to participate in the study;
* whose parent or legal guardian were perceived as unreliable or unavailable for the duration of the study period;
* who had a previous or suspected disease caused by N meningitidis;
* who had household contact with and/or intimate exposure to an individual with culture-proven N. meningitidis infection within 60 days prior to enrollment;
* who had previously been immunized with a meningococcal vaccine or vaccine containing meningococcal antigen(s) (licensed or investigational);
* who had received any investigational agents or vaccines within 90 days prior to enrollment or who expected to receive an investigational agent or vaccine prior to the completion of the study;
* who had received any licensed vaccines within one month prior to enrollment or for whom receipt of a licensed vaccine was anticipated within one month after vaccination (Exception: influenza vaccine could be administered up to 15 days prior to study vaccination and no less than 15 days after study vaccination);
* who had received a live viral vaccine within 60 days prior to enrollment;
* who had experienced, within the 7 days prior to enrollment, significant acute or chronic infection (for example requiring systemic antibiotic treatment or antiviral therapy) or had experienced fever (defined as axillary temperature ≥38°C) within 3 days prior to enrollment;
* who had any serious acute, chronic or progressive disease (e.g., any history of neoplasm, cancer, diabetes, cardiac disease, autoimmune disease, Human Immunodeficiency Virus (HIV) infection or Acquired Immune Deficiency Syndrome (AIDS), or blood dyscrasias, with signs of cardiac or renal failure or severe malnutrition). (Exception: subjects with mild asthma were eligible for enrollment; subjects with moderate or severe asthma requiring routine use of inhaled or systemic corticosteroids were not eligible for enrollment);
* who had epilepsy or any progressive neurological disease;
* who had a history of any anaphylaxis, serious vaccine reactions, or allergy to any vaccine component;
* who had a known or suspected impairment/alteration of immune function, either congenital or acquired or resulting from (for example):
* receipt of immunosuppressive therapy within 30 days prior to enrollment (any systemic corticosteroid administered for more than 5 days, or in a daily dose >1 mg/kg/day prednisone or equivalent during any of 30 days prior to enrollment, or cancer chemotherapy);
* receipt of immunostimulants;
* receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within 90 days prior to enrollment and for the full length of the study;
* common childhood exanthematous diseases (varicella, mumps, measles, rubella) occurring 6 weeks prior to vaccination;
* who were known to have a bleeding diathesis or any condition that could be associated with a prolonged bleeding time;
* who had Down syndrome or other known cytogenic disorders;
* whose families were planning to leave the area of the study site before the end of the study period;
* who had any condition that, in the opinion of the investigator, could interfere with the evaluation of the study objectives.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1500 (Actual)
Dates: Start 2006-05; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines & Diagnostics, Study Chair — Novartis Vaccines & Diagnostics
Locations (3):
- Argentina (3):
  - FUNCEI, French 3085, Buenos Aires
  - Centro di Desarrollo de Proyectos Avanzados (CEDEPAP) Roma 1464, Córdoba
  - Hospital de Pediatria "Sor Maria Ludovica", Calle 14 N1631,(1900), La Plata

REFERENCES:
- [Result] Black S, Klein NP, Shah J, Bedell L, Karsten A, Dull PM. Immunogenicity and tolerability of a quadrivalent meningococcal glycoconjugate vaccine in children 2-10 years of age. Vaccine. 2010 Jan 8;28(3):657-63. doi: 10.1016/j.vaccine.2009.10.104. Epub 2009 Nov 4. PMID 19895922

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 3 study centers in Argentina.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- MenACWY-PS: Subjects ≥2 to ≤10 years of age received one dose of a quadrivalent meningococcal polysaccharide vaccine (MenACWY-PS)
Period: Overall Study
Arm/Group | MenACWY-CRM | MenACWY-PS
Started | 950 | 550
Completed | 944 | 546
Not Completed | 6 | 4
Not completed — Withdrawal by Subject | 6 | 4

BASELINE CHARACTERISTICS:
Population: Analysis was done on all enrolled subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | MenACWY-CRM | MenACWY-PS | Total
Number analyzed (Participants) | 950 | 550 | 1500
Age, Continuous [Mean (Standard Deviation); unit: Years] | 5.8 (2.5) | 5.7 (2.5) | 5.8 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 482 | 288 | 770
  Male | 468 | 262 | 730

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With hSBA Seroresponse Against Serogroups A, C, W and Y One Month After Vaccination With MenACWY-CRM or MenACWY-PS
Description: Immunogenicity was measured as the percentage of subjects with hSBA seroresponse, directed against each of meningococcal serogroups A, C, W and Y, evaluated by serum bactericidal assay using human complement (hSBA), one month after vaccination (day 29)with MenACWY-CRM or MenACWY-PS vaccine.
  Seroresponse was defined as:
  1. for subjects with a prevaccination hSBA titer <1:4, a postvaccination hSBA titer ≥1:8;
  2. for subjects with a prevaccination hSBA titer ≥1:4, an increase in hSBA titer of at least four times the prevaccination titer.
Time Frame: 1 month after vaccination (day 29)
Population: Analysis was done on the per-protocol (PP) dataset of primary vaccination, i.e. the subjects who received the vaccine correctly; provided evaluable serum samples at one month after vaccination; and had no major protocol violations as defined in the analysis plan.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY-CRM | MenACWY-PS
Number analyzed (Participants) | 148 | 148
Percentage of subjects
  Serogroup A | 93 [87 to 96] | 55 [46 to 63]
  Serogroup C (N=147,144) | 82 [74 to 88] | 52 [44 to 60]
  Serogroup W (N=143,142) | 74 [66 to 81] | 46 [37 to 54]
  Serogroup Y (N=146,146) | 82 [74 to 87] | 63 [55 to 71]
Statistical Analysis 1: Comparison: MenACWY-CRM vs MenACWY-PS; Comparison of hSBA seroresponse for the serogroup A one month after vaccination of MenACWY-CRM and MenACWY-PS; Test type: Non-Inferiority or Equivalence — The null hypothesis was that for the serogroup A, the seroresponse percentage in the MenACWY-CRM group would be at least 10% lower than that in the MenACWY-PS group at one month postvaccination, i.e. the lower limit of the 95% CI of the difference in response rates (MenACWY-CRM minus MenACWY-PS) ≤-10%; Chi-squared; Group difference = 38, 95% CI 2-sided [29 to 47]
Statistical Analysis 2: Comparison: MenACWY-CRM vs MenACWY-PS; Comparison of hSBA seroresponse for the serogroup C one month after vaccination of MenACWY-CRM and MenACWY-PS; Test type: Non-Inferiority or Equivalence — The null hypothesis was that for the serogroup C, the seroresponse percentage in the MenACWY-CRM group would be at least 10% lower than that in the MenACWY-PS group at one month postvaccination, i.e. the lower limit of the 95% CI of the difference in response rates (MenACWY-CRM minus MenACWY-PS) ≤-10%; Chi-squared; Group difference = 30, 95% CI 2-sided [19 to 40]
Statistical Analysis 3: Comparison: MenACWY-CRM vs MenACWY-PS; Comparison of hSBA seroresponse for the serogroup W one month after vaccination of MenACWY-CRM and MenACWY-PS; Test type: Non-Inferiority or Equivalence — The null hypothesis was that for the serogroup W, the seroresponse percentage in the MenACWY-CRM group would be at least 10% lower than that in the MenACWY-PS group at one month postvaccination, i.e. the lower limit of the 95% CI of the difference in response rates (MenACWY-CRM minus MenACWY-PS) ≤-10%; Chi-squared; Group difference = 28, 95% CI 2-sided [17 to 39]
Statistical Analysis 4: Comparison: MenACWY-CRM vs MenACWY-PS; Comparison of hSBA seroresponse for the serogroup Y one month after vaccination of MenACWY-CRM and MenACWY-PS; Test type: Non-Inferiority or Equivalence — The null hypothesis was that for the serogroup Y, the seroresponse percentage in the MenACWY-CRM group would be at least 10% lower than that in the MenACWY-PS group at one month postvaccination, i.e. the lower limit of the 95% CI of the difference in response rates (MenACWY-CRM minus MenACWY-PS) ≤-10%; Chi-squared; Group difference = 18, 95% CI 2-sided [8 to 28]

2. Primary Outcome: Number of Subjects With At Least One Severe Systemic Reaction to MenACWY-CRM or MenACWY-PS Within 7 Days Postvaccination
Description: Safety was assessed in terms of the number of subjects who reported at least one severe systemic reaction after vaccination with MenACWY-CRM or MenACWY-PS from day 1 to day 7 after vaccination.
Time Frame: Day 1 to 7 postvaccination
Population: Analysis was done on the safety set, i.e. the subjects in the exposed population who provided postvaccination safety data.
Measure: Number; unit: Number of subjects
Arm/Group | MenACWY-CRM | MenACWY-PS
Number analyzed (Participants) | 950 | 550
Number of subjects | 11 | 1
Statistical Analysis 1: Comparison: MenACWY-CRM vs MenACWY-PS; Test type: Non-Inferiority or Equivalence — Safety of MenACWY-CRM vaccination was considered non-inferior to the safety of MenACWY-PS vaccination if the upper limit of the two-sided 95% CI of the ratio (MenACWY-CRM group divided by MenACWY-PS group) of the percentage of subjects experiencing at least one severe systemic reaction during 1 to 7 days after vaccination was less than 3; Risk ratio(MenACWY-CRM/MenACWY-PS); Group Ratio = 6.37, 95% CI 2-sided [0.82 to 49.2]

3. Secondary Outcome: Percentage of Subjects With hSBA Titers ≥1:4 and ≥1:8 Against Serogroups A, C, W and Y One Month After Vaccination With MenACWY-CRM or MenACWY-PS
Description: Immunogenicity was measured as the percentage of subjects who achieved hSBA titers ≥1:4 and ≥1:8 against each of four meningococcal serogroups A, C, W and Y at baseline (day 1) and one month (day 29)after one vaccination with MenACWY-CRM or MenACWY-PS.
Time Frame: Day 1 and 29
Population: Analysis was performed on the PP dataset of primary vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY-CRM | MenACWY-PS
Number analyzed (Participants) | 148 | 148
Percentage of subjects
  Serogroup A (hSBA ≥1:4)- Day 1 | 5 [2 to 10] | 3 [1 to 8]
  Serogroup A (hSBA ≥1:4)- Day 29 | 95 [90 to 98] | 55 [47 to 64]
  Serogroup C (hSBA ≥1:4)- Day 1 (N=147,144) | 26 [19 to 34] | 31 [23 to 39]
  Serogroup C (hSBA ≥1:4)- Day 29 (N=147,144) | 91 [85 to 95] | 80 [72 to 86]
  Serogroup W (hSBA ≥1:4)- Day 1 (N=143,142) | 40 [32 to 48] | 37 [29 to 46]
  Serogroup W (hSBA ≥1:4)- Day 29 (N=143,142) | 99 [96 to 100] | 78 [70 to 85]
  Serogroup Y (hSBA ≥1:4)- Day 1 (N=146,146) | 17 [11 to 24] | 15 [10 to 22]
  Serogroup Y (hSBA ≥1:4)- Day 29 (N=146,146) | 90 [84 to 95] | 77 [69 to 83]
  Serogroup A (hSBA ≥1:8)- Day 1 | 4 [2 to 9] | 2 [0 to 6]
  Serogroup A (hSBA ≥1:8)- Day 29 | 95 [90 to 98] | 55 [47 to 64]
  Serogroup C (hSBA ≥1:8)- Day 1 (N=147,144) | 16 [10 to 23] | 20 [14 to 28]
  Serogroup C (hSBA ≥1:8)- Day 29 (N=147,144) | 88 [82 to 93] | 70 [62 to 77]
  Serogroup W (hSBA ≥1:8)- Day 1 (N=143,142) | 38 [30 to 46] | 35 [27 to 43]
  Serogroup W (hSBA ≥1:8)- Day 29 (N=143,142) | 99 [96 to 100] | 73 [64 to 80]
  Serogroup Y (hSBA ≥1:8)- Day 1 (N=146,146) | 14 [9 to 21] | 11 [6 to 17]
  Serogroup Y (hSBA ≥1:8)- Day 29 (N=146,146) | 89 [83 to 94] | 66 [58 to 74]

4. Secondary Outcome: The hSBA Geometric Mean Titers Against Serogroups A, C, W and Y One Month After Vaccination With MenACWY-CRM or MenACWY-PS
Description: The immune response was measured as the hSBA geometric mean titers (GMTs) directed against each of four meningococcal serogroups A, C, W and Y at baseline (day 1) and one month(day 29) after one vaccination with MenACWY-CRM or MenACWY-PS.
Time Frame: Day 1 and 29
Population: Analysis was performed on the PP dataset of primary vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titers
Arm/Group | MenACWY-CRM | MenACWY-PS
Number analyzed (Participants) | 148 | 148
Geometric Mean Titers
  Serogroup A - Day 1 | 2.25 [2.10 to 2.41] | 2.09 [1.95 to 2.24]
  Serogroup A - Day 29 | 65 [51 to 82] | 11 [8.66 to 14]
  Serogroup C (N=147,144) - Day 1 | 3.09 [2.69 to 3.53] | 3.27 [2.85 to 3.75]
  Serogroup C (N=147,144) - Day 29 | 42 [32 to 54] | 20 [15 to 26]
  Serogroup W (N=143,142) - Day 1 | 6.22 [4.90 to 7.90] | 5.40 [4.25 to 6.87]
  Serogroup W (N=143,142) - Day 29 | 72 [56 to 92] | 20 [16 to 26]
  Serogroup Y (N=146,146) - Day 1 | 2.81 [2.48 to 3.19] | 2.64 [2.33 to 2.99]
  Serogroup Y (N=146,146) - Day 29 | 47 [35 to 63] | 25 [19 to 34]

5. Secondary Outcome: Percentage of Subjects With Persisting hSBA Titers ≥1:4 and ≥1:8 Against Serogroups A, C, W and Y at Day 181 After Vaccination With MenACWY-CRM or MenACWY-PS
Description: The persistence of immune response was measured as the percentage of subjects with hSBA titers ≥1:4 and ≥1:8 against each of four meningococcal serogroups A, C, W and Y at day 181 after vaccination with MenACWY-CRM or MenACWY-PS.
Time Frame: Day 181
Population: Analysis was performed on PP dataset for persistence analysis at day 181.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY-CRM | MenACWY-PS
Number analyzed (Participants) | 145 | 144
Percentage of subjects
  Serogroup A(≥1:4)-Day 29 (1 month postvaccination) | 96 [91 to 98] | 54 [46 to 62]
  Serogroup A(≥1:4)-Day 181(6 months postvaccination | 39 [31 to 47] | 41 [33 to 49]
  Serogroup C (hSBA ≥1:4) - Day 29 (N=141,139) | 91 [85 to 95] | 79 [71 to 86]
  Serogroup C (hSBA ≥1:4) - Day 181 (N=141,139) | 87 [81 to 92] | 71 [63 to 79]
  Serogroup W (hSBA ≥1:4) - Day 29 (N=137,137) | 99 [96 to 100] | 78 [70 to 85]
  Serogroup W (hSBA ≥1:4) - Day 181 (N=137,137) | 97 [93 to 99] | 69 [60 to 76]
  Serogroup Y (hSBA ≥1:4) - Day 29 (N=140,141) | 90 [84 to 94] | 77 [69 to 83]
  Serogroup Y (hSBA ≥1:4) - Day 181 (N=140,141) | 94 [88 to 97] | 65 [56 to 72]
  Serogroup A (hSBA ≥1:8) - Day 29 | 95 [90 to 98] | 54 [46 to 62]
  Serogroup A (hSBA ≥1:8) - Day 181 | 35 [27 to 44] | 38 [30 to 47]
  Serogroup C (hSBA ≥1:8) - Day 29 (N=141,139) | 88 [81 to 93] | 70 [61 to 77]
  Serogroup C (hSBA ≥1:8) - Day 181 (N=141,139) | 81 [73 to 87] | 55 [47 to 64]
  Serogroup W (hSBA ≥1:8) - Day 29 (N=137,137) | 99 [96 to 100] | 72 [64 to 80]
  Serogroup W (hSBA ≥1:8) - Day 181 (N=137,137) | 96 [92 to 99] | 66 [57 to 74]
  Serogroup Y (hSBA ≥1:8) - Day 29 (N=140,141) | 89 [82 to 93] | 67 [59 to 75]
  Serogroup Y (hSBA ≥1:8) - Day 181 (N=140,141) | 89 [83 to 94] | 59 [50 to 67]

6. Secondary Outcome: The hSBA Geometric Mean Titers Persisting Against Meningococcal Serogroups A, C, W and Y at Day 181 After Vaccination With MenACWY-CRM or MenACWY-PS
Description: The persistence of immune response was measured in terms of the hSBA GMTs persisting at day 181 against each of four meningococcal serogroups A, C, W and Y after vaccination with MenACWY-CRM or MenACWY-PS
Time Frame: Day 181
Population: Analysis was performed on the PP dataset for persistence analysis at day 181.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titers
Arm/Group | MenACWY-CRM | MenACWY-PS
Number analyzed (Participants) | 145 | 144
Geometric Mean Titers
  Serogroup A - Day 29 (1 month post vaccination) | 66 [52 to 83] | 11 [8.33 to 13]
  Serogroup A - Day 181 (6 months post vaccination) | 5.06 [4.05 to 6.33] | 5.85 [4.68 to 7.32]
  Serogroup C (N=141,139) - Day 29 | 41 [31 to 54] | 20 [15 to 27]
  Serogroup C (N=141,139) - Day 181 | 22 [17 to 28] | 11 [8.84 to 14]
  Serogroup W (N=137,137) - Day 29 | 74 [58 to 95] | 21 [16 to 27]
  Serogroup W (N=137,137) - Day 181 | 69 [54 to 89] | 16 [13 to 21]
  Serogroup Y (N=140,141) - Day 29 | 47 [35 to 64] | 26 [19 to 35]
  Serogroup Y (N=140,141) - Day 181 | 39 [29 to 51] | 14 [11 to 19]

7. Secondary Outcome: Number of Subjects Reporting Local and Systemic Reactions and Axillary Temperature During 7-Day Period After Vaccination With MenACWY-CRM or MenACWY-PS
Description: Safety was assessed as the number of subjects who reported local and systemic reactions and axillary temperature during day 1 to day 7 after vaccination with MenACWY-CRM or MenACWY-PS.
Time Frame: Day 1 to 7 postvaccination
Population: Analysis was performed on safety dataset. Groups were sub-divided into 2 to 5 years of age and 6 to 10 years of age.
Measure: Number; unit: participants
Groups:
- MenACWY-CRM_2 to 5 Years: Subjects ≥2 to ≤5 years of age received one vaccination of a quadrivalent meningococcal conjugate vaccine (MenACWY-CRM)
- MenACWY-PS_2 to 5 Years: Subjects ≥2 to ≤5 years of age received one vaccination of a quadrivalent meningococcal polysaccharide vaccine (MenACWY-PS)
- MenACWY-CRM_6 to 10 Years: Subjects ≥6 to ≤10 years of age received one vaccination of a quadrivalent meningococcal conjugate vaccine (MenACWY-CRM)
- MenACWY-PS_6 to 10 Years: Subjects ≥6 to ≤10 years of age received one vaccination of a quadrivalent meningococcal polysaccharide vaccine (MenACWY-PS)
Arm/Group | MenACWY-CRM_2 to 5 Years | MenACWY-PS_2 to 5 Years | MenACWY-CRM_6 to 10 Years | MenACWY-PS_6 to 10 Years
Number analyzed (Participants) | 452 | 264 | 498 | 286
participants
  Any local reaction | 138 | 99 | 189 | 125
  Injection site pain | 89 | 68 | 132 | 100
  Injection site erythema | 75 | 34 | 91 | 37
  Injection site induration | 59 | 23 | 84 | 38
  Any systemic reaction | 130 | 73 | 119 | 69
  Change in Eating Habits | 36 | 24 | NA — This systemic reaction is not applicable to this age group | NA — This systemic reaction is not applicable to this age group
  Sleepiness | 29 | 13 | NA — This systemic reaction is not applicable to this age group | NA — This systemic reaction is not applicable to this age group
  Irritability | 36 | 18 | NA — This systemic reaction is not applicable to this age group | NA — This systemic reaction is not applicable to this age group
  Vomiting | 21 | 9 | NA — This systemic reaction is not applicable to this age group | NA — This systemic reaction is not applicable to this age group
  Diarrhea | 31 | 20 | NA — This systemic reaction is not applicable to this age group | NA — This systemic reaction is not applicable to this age group
  Arthralgia | 26 | 11 | 18 | 15
  Headache | 46 | 22 | 74 | 46
  Chills | NA — This systemic reaction is not applicable to this age group | NA — This systemic reaction is not applicable to this age group | 18 | 17
  Nausea | NA — This systemic reaction is not applicable to this age group | NA — This systemic reaction is not applicable to this age group | 16 | 11
  Malaise | NA — This systemic reaction is not applicable to this age group | NA — This systemic reaction is not applicable to this age group | 50 | 28
  Myalgia | NA — This systemic reaction is not applicable to this age group | NA — This systemic reaction is not applicable to this age group | 35 | 25
  Any other AE | 69 | 42 | 69 | 47
  Axillary Temperature ≥38 °C | 35 | 18 | 20 | 16
  Analgesic/Antipyretic medicine used | 69 | 42 | 69 | 47

ADVERSE EVENTS:
Time Frame: Solicited adverse events (AEs) were collected from Day 1 through 7,Serious AEs were collected from day 1 to day 181 after vaccination.
Arm/Group | MenACWY-CRM | MenACWY-PS
Serious Adverse Events (participants affected / at risk) | 9/950 | 1/550
Other Adverse Events (participants affected / at risk) | 409/950 | 271/550
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACWY-CRM (N=950) | MenACWY-PS (N=550)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Lobar Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Febrile Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Tonic Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Asthmatic Crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACWY-CRM (N=950) | MenACWY-PS (N=550)
Injection site pain (General disorders) | 221 (221) | 168 (168)
Injection site erythema (General disorders) | 166 (166) | 71 (71)
Headache (Nervous system disorders) | 125 (125) | 72 (72)
Injection site induration (General disorders) | 143 (143) | 61 (61)
Pyrexia (General disorders) | 75 (75) | 49 (49)
Malaise (General disorders) | 50 (50) | 28 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days